CLINICAL TRIAL: NCT06820957
Title: Randomized Phase 2/3 Trial of Vincristine-Irinotecan-Regorafenib in Combination With Vincristine-Doxorubicin-Cyclophosphamide (VDC) and Ifosfamide-Etoposide (IE) in Patients With Newly Diagnosed Metastatic Ewing Sarcoma
Brief Title: Testing a New Combination of Anti-cancer Drugs in Patients Newly Diagnosed With Ewing Sarcoma Who Have Cancer That Has Spread to Other Parts of the Body
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AEWS2431; NCI-2025-00801 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); AEWS2431 (Other: Children's Oncology Group); AEWS2431 (Other: CTEP); U10CA180886 (NIH)
Record Dates: First submitted 2025-02-06; First posted 2025-02-11 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: CIC-Rearranged Sarcoma; Metastatic Ewing Sarcoma; Metastatic High Grade Sarcoma; Metastatic Undifferentiated Round Cell Sarcoma; Metastatic Undifferentiated Sarcoma, Not Otherwise Specified; Round Cell Sarcoma With EWSR1-non-ETS Fusion; Sarcoma With BCOR Genetic Alterations
MeSH Terms: conditions — Sarcoma, Ewing | interventions — Biopsy; Specimen Handling; Cyclophosphamide; Doxorubicin; Etoposide; Fluorodeoxyglucose F18; Ifosfamide; Irinotecan; Magnetic Resonance Spectroscopy; Radiotherapy; Radiation; regorafenib; Surgical Procedures, Operative; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Regimen A (VDC/IE) (Active Comparator): See Detailed description
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Procedure: Computed Tomography; Drug: Cyclophosphamide; Drug: Doxorubicin Hydrochloride; Procedure: Echocardiography Test; Drug: Etoposide; Other: Fludeoxyglucose F-18; Drug: Ifosfamide; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography; Other: Questionnaire Administration; Radiation: Radiation Therapy; Procedure: Surgical Procedure; Drug: Vincristine Sulfate
- Regimen B (VIrR/VDC/IE) (Experimental): See Detailed Description
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Procedure: Computed Tomography; Drug: Cyclophosphamide; Drug: Doxorubicin Hydrochloride; Procedure: Echocardiography Test; Drug: Etoposide; Other: Fludeoxyglucose F-18; Drug: Ifosfamide; Drug: Irinotecan Hydrochloride; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography; Other: Questionnaire Administration; Radiation: Radiation Therapy; Drug: Regorafenib; Procedure: Surgical Procedure; Drug: Vincristine Sulfate

INTERVENTIONS:
Procedure: Biopsy Procedure — Undergo bone marrow aspiration and biopsy
  Other Names: Biopsy; BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo tissue and/or blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Marrow Aspiration — Undergo bone marrow aspiration and biopsy
Procedure: Bone Marrow Biopsy — Undergo bone marrow aspiration and biopsy
  Other Names: Biopsy of Bone Marrow; Biopsy, Bone Marrow
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Asta B 518; B 518; B-518; B518; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR 138719; WR- 138719; WR-138719; WR138719
Drug: Doxorubicin Hydrochloride — Given IV
  Other Names: 5,12-Naphthacenedione, 10-[(3-amino-2,3,6-trideoxy-alpha-L-lyxo-hexopyranosyl)oxy]-7,8, 9,10-tetrahydro-6,8,11-trihydroxy-8-(hydroxyacetyl)-1-methoxy-, hydrochloride, (8S-cis)- (9CI); ADM; Adriacin; Adriamycin; Adriamycin Hydrochloride; Adriamycin PFS; Adriamycin RDF; ADRIAMYCIN, HYDROCHLORIDE; Adriamycine; Adriblastina; Adriblastine; Adrimedac; Chloridrato de Doxorrubicina; DOX; DOXO-CELL; Doxolem; Doxorubicin HCl; Doxorubicin.HCl; Doxorubin; Farmiblastina; FI 106; FI-106; FI106; hydroxydaunorubicin; Rubex
Procedure: Echocardiography Test — Undergo echocardiography
  Other Names: EC; Echocardiography
Drug: Etoposide — Given IV
  Other Names: Demethyl Epipodophyllotoxin Ethylidine Glucoside; EPEG; Lastet; Toposar; Vepesid; VP 16; VP 16-213; VP 16213; VP-16; VP-16-213; VP-16213; VP16; VP16213
Other: Fludeoxyglucose F-18 — Given FDG
  Other Names: 18FDG; FDG; Fludeoxyglucose (18F); fludeoxyglucose F 18; Fludeoxyglucose F18; Fluorine-18 2-Fluoro-2-deoxy-D-Glucose; Fluorodeoxyglucose F18
Drug: Ifosfamide — Given IV
  Other Names: Asta Z 4942; Asta Z-4942; Cyfos; Holoxan; Holoxane; Ifex; IFO; IFO-Cell; Ifolem; Ifomida; Ifomide; Ifosfamidum; Ifoxan; IFX; Iphosphamid; Iphosphamide; Iso-Endoxan; Isoendoxan; Isophosphamide; Mitoxana; MJF 9325; MJF-9325; Naxamide; Seromida; Tronoxal; Z 4942; Z-4942
Drug: Irinotecan Hydrochloride — Given IV
  Other Names: Campto; Camptosar; Camptothecin 11; Camptothecin-11; CPT 11; CPT-11; CPT11; Irinomedac; Irinotecan Hydrochloride Trihydrate; Irinotecan Monohydrochloride Trihydrate; U 101440E; U-101440E; U101440E
  Arms: Regimen B (VIrR/VDC/IE)
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Procedure: Positron Emission Tomography — Undergo FDG PET
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; PT
Other: Questionnaire Administration — Ancillary studies
Radiation: Radiation Therapy — Undergo radiation
  Other Names: Cancer Radiotherapy; Energy Type; ENERGY_TYPE; Irradiate; Irradiated; Irradiation; Radiation; Radiation Therapy, NOS; Radiotherapeutics; Radiotherapy; RT; Therapy, Radiation
Drug: Regorafenib — Given PO
  Other Names: BAY 73-4506 Monohydrate; BAY-73-4506 Monohydrate; Regorafenib Monohydrate; Stivarga
  Arms: Regimen B (VIrR/VDC/IE)
Procedure: Surgical Procedure — Undergo surgery
  Other Names: Operation; Surgery; Surgery Type; Surgery, NOS; Surgical; Surgical Intervention; Surgical Interventions; Surgical Procedures; Type of Surgery
Drug: Vincristine Sulfate — Given IV
  Other Names: Kyocristine; Leurocristine Sulfate; Leurocristine, sulfate; Oncovin; Vincasar; Vincosid; Vincrex; Vincristine, sulfate

SUMMARY:
This phase II/III trial compares the effect of vincristine, irinotecan, and regorafenib (VIrR) in combination with vincristine, doxorubicin, cyclophosphamide (VDC), ifosfamide and etoposide (IE) to usual treatment with VDC/IE for the treatment of newly diagnosed Ewing sarcoma or other round cell sarcomas that have spread from where they first started (primary site) to other places in the body (metastatic). Vincristine is in a class of medications called vinca alkaloids. It works by stopping tumor cells from growing and dividing and may kill them. Irinotecan is in a class of antineoplastic medications called topoisomerase I inhibitors. It blocks a certain enzyme needed for cell division and deoxyribonucleic acid (DNA) repair and may kill tumor cells. Regorafenib, a type of kinase inhibitor and a type of antiangiogenesis agent, blocks certain proteins, which may help keep tumor cells from growing. It may also prevent the growth of new blood vessels that tumors need to grow. Doxorubicin is in a class of medications called anthracyclines. Doxorubicin damages the cell's DNA and may kill tumor cells. It also blocks a certain enzyme needed for cell division and DNA repair. Cyclophosphamide is in a class of medications called alkylating agents. It works by damaging the cell's DNA and may kill tumor cells. It may also lower the body's immune response. Ifosfamide, a type of alkylating agent and a type of antimetabolite, attaches to DNA in cells and may kill tumor cells. Etoposide is in a class of medications known as podophyllotoxin derivatives. It blocks a certain enzyme needed for cell division and DNA repair and may kill tumor cells. Giving VIrR/VDC/IE may be more effective than usual treatment with VDC/IE in treating patients with newly diagnosed metastatic Ewing sarcoma or other round cell sarcomas.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine if the event-free survival (EFS) in patients with newly diagnosed metastatic Ewing sarcoma is improved when treated with vincristine-irinotecan-regorafenib (VIrR) after initial treatment with vincristine-doxorubicin-cyclophosphamide (VDC) and ifosfamide-etoposide (IE) compared to patients treated with 17 cycles of interval compressed VDC and IE chemotherapy.

SECONDARY OBJECTIVES:

I. To compare the overall survival (OS) of patients with newly diagnosed metastatic Ewing sarcoma treated with VDC/IE/VIrR versus VDC/IE.

II. To compare the toxicity profile of VDC/IE/VIrR to VDC/IE in patients with newly diagnosed metastatic Ewing sarcoma, using both investigator-reported and patient-reported Common Terminology Criteria for Adverse Events (CTCAE).

III. To describe the feasibility and toxicity of augmented dose radiotherapy with 64.8 Gy as local control for patients with newly diagnosed metastatic Ewing sarcoma with large primary tumors.

IV. To prospectively validate that circulating tumor-derived DNA (ctDNA) levels greater than or equal to 5% at the time of diagnosis are associated with increased risk of EFS-event for patients with newly diagnosed metastatic Ewing sarcoma.

V. To prospectively validate that elevated ctDNA levels greater than or equal to 0.5% burden following one cycle of chemotherapy are associated with increased risk of EFS-event for patients with newly diagnosed metastatic Ewing sarcoma.

EXPLORATORY OBJECTIVES:

I. To estimate 1- and 2-year EFS and response rate for patients with newly diagnosed, eligible metastatic round cell sarcomas other than Ewing sarcoma.

II. To characterize the change in fludeoxyglucose F-18 (FDG)-positron emission tomography (PET) imaging response of primary disease site at the end of Induction chemotherapy and its association with EFS.

III. To explore distinguishing histologic attributes of Ewing sarcoma and round cell sarcomas that mimic Ewing sarcoma.

IV. To collect bone marrow and tissue samples to bank for future research. V. To explore other ctDNA predictor variables, time points, and potential association with EFS in patients with newly diagnosed metastatic Ewing sarcoma.

VI. To estimate the frequency of selected toxicities by Patient Reported Outcomes (PRO)-CTCAE and symptom bother by Functional Assessment of Cancer Therapy General Questionnaire (FACT-G) and to evaluate if these findings are associated with duration of protocol therapy and treatment arm.

OUTLINE:

INDUCTION: Patients receive vincristine intravenously (IV) on days 1 and 8, doxorubicin IV over 3-15 minutes on days 1 and 2, and cyclophosphamide IV over 30-60 minutes on day 1 of cycles 1, 3 and 5. Patients also receive ifosfamide IV over 1 hour and etoposide IV over 1 hour on days 1-5 of cycles 2, 4 and 6. Cycles repeat every 14 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Patients then undergo surgery or radiation therapy per investigator choice.

CONSOLIDATION I: Patients receive vincristine IV on days 1 and 8, doxorubicin IV over 3-15 minutes on days 1 and 2, and cyclophosphamide IV over 30-60 minutes on day 1 of cycles 1 and 2. Patients also receive ifosfamide IV over 1 hour and etoposide IV over 1 hour on days 1-5 of cycles 3 and 4. Cycles repeat every 14 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity.

CONSOLIDATION II: After 10 cycles of therapy, patients with Ewing Sarcoma are randomized to 1 of 2 regimens. Patients with a diagnosis of other eligible metastatic round cell sarcomas are assigned to Regimen A.

REGIMEN A: Patients receive vincristine IV on days 1 and 8 and cyclophosphamide IV over 30-60 minutes on day 1 of cycles 1, 3, 5 and 7. Patients also receive ifosfamide IV over 1 hour and etoposide IV over 1 hour on days 1-5 of cycles 2, 4 and 6. Cycles repeat every 14 days for up to 7 cycles in the absence of disease progression or unacceptable toxicity. After systemic therapy completed, patients undergo metastatic site radiation therapy.

REGIMEN B: Patients receive vincristine IV on days 1 and 8 and irinotecan IV over 90 minutes on days 1-5 of each cycle. Patients also receive regorafenib orally (PO) on days 8-14 or 15-21 of cycle 1, and then on days 8-21 of cycles thereafter. Cycles repeat every 21 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity. After systemic therapy completed, patients undergo metastatic site radiation therapy.

Additionally, patients undergo blood sample collection, echocardiography, magnetic resonance imaging (MRI), computed tomography (CT), chest CT, and/or FDG-PET throughout the study. Patients may also undergo optional collection of tumor tissue and/or bone marrow aspiration and biopsy on study.

After completion of study treatment, patients are followed every 3 months for years 1 and 2, every 6 months for years 3 and 4 then every 12 months for years 5-10.

ELIGIBILITY:
Inclusion Criteria:

* All patients must be enrolled on APEC14B1 and consented to the Molecular Characterization Initiative (Part A) prior to enrollment and treatment on AEWS2431
* Patients must be ≥ 12 months to ≤ 50 years of age at time of enrollment
* Newly diagnosed Ewing sarcoma and other round cell sarcomas as follows. For the purposes of eligibility, the following pathology diagnoses are eligible and molecular confirmation is not required to enroll:

  * Histologically confirmed Ewing sarcoma
  * Suspected Ewing sarcoma with molecular confirmation pending
  * Suspected high grade round cell sarcomas/sarcomas with eligible molecular alterations, pending molecular confirmation
  * Round cell sarcoma consistent with Ewing sarcoma
  * Round cell sarcoma not otherwise specified
  * Round cell sarcoma
  * Round cell sarcomas with EWSR1-non-ETS fusion
  * CIC-rearranged sarcoma
  * Sarcoma with BCOR genetic alterations
* Patients with the following pathologic diagnoses that are known to contain EWSR1 or FUS fusions are not eligible:

  * Angiomatoid fibrous histiocytoma
  * Extraskeletal myxoid chondrosarcoma
  * Desmoplastic small round cell tumor
  * Clear cell sarcoma
  * Myxoid liposarcoma
* If clinical molecular testing that reports both fusion partners has been successfully completed by the site prior to enrollment, patients may only enroll if that testing reported one of the eligible fusions
* All patients must have evidence of distant metastatic disease. Biopsy of metastatic sites is not required. For this study, distant metastatic disease is defined as one or more of the following:

  * Lesions which are discontinuous from the primary tumor, are not regional lymph nodes, and do not share a bone or body cavity with the primary tumor. Skip lesions in the same bone as the primary tumor do not constitute metastatic disease. Skip lesions in an adjacent bone are considered bone metastasis. If there is any doubt whether lesions are metastatic, a biopsy of those lesions should be performed
  * Contralateral pleural effusion and/or contralateral pleural nodules
  * Distant lymph node involvement
  * Patients with pulmonary nodules are considered to have metastatic disease if the patient has:

    * Solitary nodule ≥ 0.5 cm or multiple nodules of ≥ 0.3 cm unless lesion is biopsied and negative for tumor
    * Patients with solitary nodule < 0.5 cm or multiple nodules < 0.3 cm are not considered to have lung metastasis unless biopsy documents tumor
  * Bone marrow metastatic disease (bone marrow disease) is based on morphologic evidence of Ewing sarcoma based on hematoxylin and eosin (H&E) stains. In the absence of morphologic evidence of marrow involvement on H&E, patients with bone marrow involvement detected ONLY by flow cytometry, reverse transcriptase-polymerase chain reaction (RT-PCR), fluorescence in situ hybridization (FISH), immunohistochemistry or PET-CT will NOT be considered to have clinical bone marrow involvement for the purposes of this study
* Creatinine clearance or radioisotope glomerular filtration rate (GFR) ≥ 50 mL/min/1.73 m^2 or serum creatinine based on age/sex as follows:

  * Age: 1 to < 2 years: Male 0.6; female 0.6
  * Age: 2 to < 6 years: Male 0.8; female 0.8
  * Age: 6 to < 10 years: Male 1; female 1
  * Age: 10 to < 13 years: Male 1.2; female 1.2
  * Age: 13 to < 16 years: Male 1.5; female 1.4
  * Age: ≥ 16 years: Male 1.7; female 1.4 OR
  * A 24-hour urine creatinine clearance ≥ 50 mL/min/1.73 m^2 OR
  * A GFR ≥ 50 mL/min/1.73 m^2. GFR must be performed using direct measurement with a nuclear blood sampling method OR direct small molecule clearance method (iothalamate or other molecule per institutional standard)
* Total bilirubin ≤ 1.5 x upper limit of normal (ULN) for age
* Serum glutamic pyruvic transaminase (SGPT) (alanine aminotransferase [ALT]) ≤ 3 x ULN for age (except for patients with liver metastasis who may enroll if ALT ≤ 5 times ULN for age)

  * Note: For the purpose of this study, the ULN for SGPT (ALT) has been set to the value of 45 U/L
* Shortening fraction of ≥ 27% by echocardiogram, or ejection fraction of ≥ 50% by echocardiogram
* No known congenital QT syndrome
* No known family history of congenital QT syndrome
* Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients should be class II or better
* Known HIV-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial

Exclusion Criteria:

* Patients with regional node involvement as their only site of disease beyond the primary tumor
* Patients whose primary tumors arise in the intra-dural soft tissue (e.g., brain and spinal cord)

  * Note: metastatic disease is allowable
* Patients with known Charcot-Marie-Tooth disease
* Patients who have had complete or partial resection of the primary tumor at initial diagnosis will only be eligible if adequate imaging (CT or MRI for most primary tumor sites) was obtained prior to surgery
* Patients who have received prior chemotherapy for current diagnosis, except for patients who have started cycle 1 VDC post-consent and within the timelines allowed for
* Patients who have received prior radiation therapy for current diagnosis
* Patients previously treated with a multitargeted tyrosine kinase inhibitor
* History of organ allograft (including allogeneic bone marrow transplant)
* Known hypersensitivity to regorafenib
* Active or chronic hepatitis B or C, or chronic hepatitis B or C requiring treatment with antiviral therapy
* Patients receiving strong CYP3A4 inducers or strong CYP3A4 inhibitors
* Female patients who are pregnant since fetal toxicities and teratogenic effects have been noted for several of the study drugs. A pregnancy test is required for female patients of childbearing potential
* Lactating females who plan to breastfeed their infants
* Females of childbearing potential must agree to either practice medically accepted highly-effective methods of contraception or abstain from heterosexual intercourse for the duration of the protocol therapy through 12 months after the last dose of cyclophosphamide or ifosfamide, 6 months after the last dose of doxorubicin, etoposide, and irinotecan, and 7 months after the last dose of regorafenib, whichever is longer
* Male patients with female partners of childbearing potential must agree to either practice a medically accepted highly-effective methods of contraception or abstain from heterosexual intercourse for the duration of the protocol therapy through 6 months after the last dose of doxorubicin and ifosfamide, 4 months after the last dose of cyclophosphamide, etoposide and regorafenib, and 3 months after the last dose of irinotecan, whichever is longer
* All patients and/or their parents or legal guardians must sign a written informed consent
* All institutional, Food and Drug Administration (FDA), and National Cancer Institute (NCI) requirements for human studies must be met

Ages: 12 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 437 (Estimated)
Dates: Start 2025-11-10 (Actual); Primary Completion 2032-07-15 (Estimated); Study Completion 2032-07-15 (Estimated)

PRIMARY OUTCOMES:
Time to event-free survival (EFS) post-Consolidation I (C1) | From randomization to progression or relapse, diagnosis of a second malignant neoplasm, death, or last patient contact, whichever occurs first, assessed up to 10 years
  Analysis will be done by associating each patient's outcome with the individual's randomized treatment assignment. The associated statistical tests will be stratified according to grouping.

SECONDARY OUTCOMES:
Overall survival-C1 | From randomization to death or last patient contact, whichever occurs first, assessed up to 10 years
  The stratified one-sided logrank test will be the primary statistical methodology for assessing the null statistical hypothesis.
EFS | From enrollment to progression or relapse, diagnosis of a second malignant neoplasm, death, or last patient contact, whichever occurs first, assessed up to 10 years
Incidence of adverse events (AEs) | Up to 30 days after last dose of study treatment
  Toxicity will be coded according to the Common Terminology Criteria for Adverse Events (CTCAE) version (v) 5.
Feasibility of augmented dose radiotherapy (ADRT) as local control | Up to point of radiation therapy (RT) termination
  The actual RT delivered will be compared with the treatment plan until the point of RT termination as assessed by central review. Will consider ADRT to be feasible to deliver if there is evidence that the patient-specific probability of feasibility-failure is less than 15%.
Toxicity of ADRT as local control | Up to 30 days after ADRT is completed
  Will be evaluated using CTCAE v 5.
Validation of circulating tumor-derived deoxyribonucleic acid (ctDNA) levels greater than or equal to 5% at the time of diagnosis are associated with increased risk of EFS-event | At time of diagnosis
Validation of ctDNA burden associated with increased risk of EFS-event | Following one cycle of chemotherapy at induction (cycle length = 14 days)
  Will compare the risk for EFS-event from enrollment for groups of patients defined by percent ctDNA using a two-sided logrank test.

OTHER OUTCOMES:
EFS and response rate | At 1 and 2 years
  The 95% confidence bounds will be calculated according to the complementary log-log transformation. Will report the 1-, 2- and 3-year estimate EFS probabilities as well as the confidence intervals.
Change in fludeoxyglucose F-18 positron emission tomography imaging response of primary disease site and its association with EFS | At the end of 6 cycles of induction chemotherapy (cycle length = 14 days)
  Will calculate the percent change in standardized uptake value (SUV). Will fit a Cox proportional hazards regression model for hazard of EFS-event with percent change in SUV included as an independent variable. Nonlinearity will be formally tested using a two degree of freedom Wald test of size 0.05 for the null hypothesis. The functional form of the relationship between hazard of EFS-event and percent change in SUV will be explored by plotting the model-predicted hazard on the logarithmic scale against percent change in SUV with 95% confidence bands. This plot will be examined for natural inflection points in the curve representing potentially informative categories of percent change in SUV. If the p-value for this test is not significant at the 0.05 level, will remove the nonlinear spline terms refitting the model with linear percent change in SUV, and will report the associated hazard ratio and 95% confidence interval.
Histologic attributes of Ewing sarcoma and round cell sarcomas that mimic Ewing sarcoma | Up to 10 years
  Qualitative characteristics will be quantified with the observed proportion in each category and the associated confidence interval. The sample mean, median, standard deviation, 25th percentile and 75th percentile will be used to characterize the distribution of the quantitative characteristics.
ctDNA predictor variables, time points, and potential association with EFS | Up to 10 years
Frequency of selected toxicities | Up to 12 months after completion of systemic therapy
  Will be evaluated using the Patient Reported Outcomes Version of Common Terminology Criteria for Adverse Events and Functional Assessment of Cancer Therapy General Questionnaire.
Probability of radiation recall AEs | Up to 30 days after RT is completed
  The probability of radiation recall AEs will be compared. The reporting period characteristics are indicator variables including the randomized regimen as well as the tumor sites radiated. The null hypothesis will be tested using a one-sided test against the alternative that the experimental regimen has an increased frequency of toxicity-events each time the study progress report is prepared for this trial.
Rate of refusal of randomization | Up to 10 years
Clinically Significant Treatment Modification Probability | Up to 10 years
  The null hypothesis will be tested using a one-sided test against the alternative that the experimental regimen has an increased frequency of treatment modification-events after the twentieth patient is randomized to Regimen B (or the first study progress report is due, whichever occurs first) and each time the study progress report is prepared for this trial.

CONTACTS AND LOCATIONS:
Overall Officials: Bhuvana A Setty, Principal Investigator — Children's Oncology Group
Locations (9):
- United States (9):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - Saint Jude Midwest Affiliate, Peoria, Illinois
  - NYU Langone Hospital - Long Island, Mineola, New York
  - Saint Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Prisma Health Richland Hospital, Columbia, South Carolina
  - BI-LO Charities Children's Cancer Center, Greenville, South Carolina
  - East Tennessee Childrens Hospital, Knoxville, Tennessee